CLINICAL TRIAL: NCT05870410
Title: Evaluation Of Non Infectious Warning Signs Of Inborn Errors Of Immunity In Children At Sohag University Hospital
Brief Title: Evaluation Of Non Infectious Presentation of Inborn Errors Of Immunity
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Amany Mansour Shalby, pediateric resident, Sohag University
Other Study IDs: Soh-Med-23-04-04MS
Record Dates: First submitted 2023-04-30; First posted 2023-05-23 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Inborn Errors of Immunity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Inborn errors of immunity (IEI) are a wide number of conditions featured by impaired immune response, and their classification is in a continuous update, with the discovery of new clinical entities . Historically, the warning signs to identify children at risk of IEI have been defined according to the susceptibility to multiple or severe infectious diseases. High recurrence of infections, severe infections with need for hospitalization, use of intravenous antibiotics, and delayed resolution (and recently, infections by unusual pathogens or restricted pathogen susceptibility) are universally recognized as "red flags" for IEI . Recent advances in the clinical comprehension of IEI,.

the immune dysregulation observed in patients with IEI is clinically expressed with autoimmunity, atopy, and lymphoproliferation, and these manifestations represent the first sign of the disease in about 10% of the patients .

DETAILED DESCRIPTION:
Inborn errors of immunity (IEI) are a wide number of conditions featured by impaired immune response, and their classification is in a continuous update, with the discovery of new clinical entities (1). Historically, the warning signs to identify children at risk of IEI have been defined according to the susceptibility to multiple or severe infectious diseases. High recurrence of infections, severe infections with need for hospitalization, use of intravenous antibiotics, and delayed resolution (and recently, infections by unusual pathogens or restricted pathogen susceptibility) are universally recognized as "red flags" for IEI . Recent advances in the clinical comprehension of IEI, together with the expansion of their genetic background and the formulation of specific genotype-phenotype correlations, allowed the better characterization of the non-infectious manifestations of IEI Specifically, the immune dysregulation observed in patients with IEI is clinically expressed with autoimmunity, atopy, and lymphoproliferation, and these manifestations represent the first sign of the disease in about 10% of the patients. Additionally, new diseases with predominant immune dysregulation phenotype in absence of a significant increase of infections have been identified, leading to an extension of the paradigm of immunodeficiency During the diagnostic work-up, patients with non-infectious onset of IEI are frequently addressed to different specialists, including hematologists, endocrinologists, rheumatologists, and allergologists, often resulting in a delayed diagnosis. In this paper, we provide a brief review on the non-infectious manifestations of IEI potentially evidenced at disease onset, focusing on the specific items to be considered for the different clinical specialists

ELIGIBILITY:
Inclusion Criteria:

* Children age from zero day to 18 yrs.

  * Children suffering from autoimmune cytopenia, eczema, nonmalignant lymphoproliferative disorder, autoimmune endocrinopathy, autoimmune enteropathy, rheumatological disease (SLE, vasculitis).
  * Children with positive family history for inborn error of immunity

Exclusion Criteria:

* • Children with secondary immune deficiency.

  * Persons above 18 years old.
  * Children who start therapy

Ages: 1 Day to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: - Children age from zero day to 18 yrs.
  * Children suffering from autoimmune cytopenia, eczema, nonmalignant lymphoproliferative disorder, autoimmune endocrinopathy, autoimmune enteropathy, rheumatological disease (SLE, vasculitis).
  * Children with positive family history for inborn error of immunit
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
measurement of percentage of inborn errors of immunity among screened children. | 1month
  measurement of percentage of inborn errors of immunity among screened children who presented with autoimmune cytopenia, eczema, nonmalignant lymphoproliferative disorder, autoimmune endocrinopathy, autoimmune enteropathy, rheumatological disease (SLE, vasculitis).

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tangye SG, Al-Herz W, Bousfiha A, Chatila T, Cunningham-Rundles C, Etzioni A, Franco JL, Holland SM, Klein C, Morio T, Ochs HD, Oksenhendler E, Picard C, Puck J, Torgerson TR, Casanova JL, Sullivan KE. Human Inborn Errors of Immunity: 2019 Update on the Classification from the International Union of Immunological Societies Expert Committee. J Clin Immunol. 2020 Jan;40(1):24-64. doi: 10.1007/s10875-019-00737-x. Epub 2020 Jan 17. PMID 31953710
- [Background] Giardino G, Gallo V, Prencipe R, Gaudino G, Romano R, De Cataldis M, Lorello P, Palamaro L, Di Giacomo C, Capalbo D, Cirillo E, D'Assante R, Pignata C. Unbalanced Immune System: Immunodeficiencies and Autoimmunity. Front Pediatr. 2016 Oct 6;4:107. doi: 10.3389/fped.2016.00107. eCollection 2016. PMID 27766253
- [Background] Arkwright PD, Gennery AR. Ten warning signs of primary immunodeficiency: a new paradigm is needed for the 21st century. Ann N Y Acad Sci. 2011 Nov;1238:7-14. doi: 10.1111/j.1749-6632.2011.06206.x. PMID 22129048
- [Background] Thalhammer J, Kindle G, Nieters A, Rusch S, Seppanen MRJ, Fischer A, Grimbacher B, Edgar D, Buckland M, Mahlaoui N, Ehl S; European Society for Immunodeficiencies Registry Working Party. Initial presenting manifestations in 16,486 patients with inborn errors of immunity include infections and noninfectious manifestations. J Allergy Clin Immunol. 2021 Nov;148(5):1332-1341.e5. doi: 10.1016/j.jaci.2021.04.015. Epub 2021 Apr 23. PMID 33895260